CLINICAL TRIAL: NCT04267887
Title: Advanced ChemoHormonal Therapy for Treatment Naïve Metastatic Prostate Cancer: Apalutamide and Abiraterone Acetate With Prednisone and Androgen Deprivation Therapy After Treatment With Docetaxel and Androgen Deprivation Therapy
Brief Title: Advanced ChemoHormonal Therapy for Treatment Naive Metastatic Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Julie Graff, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00016728; NCI-2020-00598 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00016728 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Castration-Sensitive Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Androgen Antagonists; apalutamide; Prednisone; deltacortene; prednylidene; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (apalutamide, abiraterone acetate, prednisone, ADT) (Experimental): Patients receive apalutamide PO QD, abiraterone acetate PO QD, and prednisone PO QD. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive androgen deprivation therapy per standard of care. Patients undergo CT scan, bone scan and blood sample collection throughout the study.
  Interventions: Drug: Abiraterone Acetate; Drug: Antiandrogen Therapy; Drug: Apalutamide; Drug: Prednisone; Procedure: Computed Tomography; Procedure: Bone Scan; Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Abiraterone Acetate — Given PO
  Other Names: CB7630; Yonsa; Zytiga
Drug: Antiandrogen Therapy — Given ADT per standard of care
  Other Names: ADT; Androgen Deprivation Therapy; Androgen Deprivation Therapy (ADT); Anti-androgen Therapy; Anti-androgen Treatment; Antiandrogen Treatment; Hormone Deprivation Therapy; Hormone-Deprivation Therapy
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; Erleada; JNJ 56021927; JNJ-56021927
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well the combination of apalutamide, abiraterone acetate, and prednisone after chemotherapy work in treating patients that have received no prior treatment (treatment naive) for high risk prostate cancer that is sensitive to androgen deprivation therapy (castration sensitive) and has spread to other parts of the body (metastatic). This study also aims to understand the inheritance of prostate cancer. If a gene or genes that cause prostate cancer can be found, the diagnosis and treatment of prostate cancer may be improved. Testosterone (a male hormone) can cause the growth of prostate cancer cells. Hormone therapy using apalutamide may fight prostate cancer by blocking the use of testosterone by the tumor cells. Antihormone therapy, such as abiraterone acetate, may lessen the amount of testosterone made by the body. Anti-inflammatory drugs such as prednisone lower the body's immune response and are used with other drugs in the treatment of some types of cancer. Apalutamide, abiraterone acetate, and prednisone after chemotherapy may work better in treating patients with castration sensitive prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Efficacy of apalutamide in combination with abiraterone acetate + prednisone following docetaxel with ongoing androgen deprivation therapy in men with high risk metastatic castration sensitive disease.

SECONDARY OBJECTIVES:

I. Safety and tolerability of apalutamide in combination with abiraterone acetate + prednisone following docetaxel with ongoing androgen deprivation therapy.

II. Time to event.

III. Depth of prostate specific antigen (PSA) response.

EXPLORATORY OBJECTIVES:

I. Quality of life.

II. Falls.

III. Molecular changes from prostate cancer over time.

OUTLINE:

Patients receive apalutamide orally (PO) once daily (QD), abiraterone acetate PO QD, and prednisone PO QD. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive androgen deprivation therapy per standard of care. Patients undergo computed tomography (CT) scan, bone scan and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 6 months for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed prostate cancer OR a strong suspicion of prostate cancer as evidenced by metastatic disease in a pattern consistent with prostate cancer (such as blastic lesions on a nuclear medicine bone scan or lymphadenopathy on the computed tomography [CT] scan) AND a PSA > 50 ng/mL
* Patients must meet either of the definitions for high risk disease as follows:

  * Definition 1: Must have at least 2 of the following 3 at the time diagnosed metastatic:

    * visceral metastatic disease
    * >=3 bone lesions
    * Gleason 8-10 OR
  * Definition 2: >=4 bone lesions, including >=1 outside of the vertebral column or pelvis and/or visceral metastatic disease
* If a patient has received androgen deprivation therapy (ADT) for neoadjuvant or adjuvant therapy at least 24 months MUST have elapsed since its use to day 1 of restarting ADT for metastatic castration sensitive disease
* ADT sensitive disease- no evidence of PSA progression or new metastatic deposits since starting ADT; PSA progression is defined as an increase in PSA greater than 25% above nadir, and >2 ng/ml increase confirmed by a second value obtained at least 2 weeks apart
* Have completed up to 6 cycles of docetaxel since developing metastatic castration sensitive disease with no more than 16 weeks elapsed since day 21 of the final cycle
* All races and ethnic groups will be included
* Life expectancy of greater than 18 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Hemoglobin > 9.0 g/dL, independent of transfusion and/or growth factors
* Leukocytes > 3,000/uL
* Absolute neutrophil count > 1,500/uL
* Platelets >= 100,000 x 10^9/uL, independent of transfusion and/or growth factors
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (Note: In subjects with Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is =< 1.5 x ULN, subject may be eligible)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) < 2.5 x institutional upper limit of normal
* Albumin > 3 g/dL
* Estimated glomerular filtration rate (eGFR) > 30 mL/min/1.73 m^2; per Modification of Diet in Renal Disease (MDRD) calculation or institutional standard
* Potassium >= 3.5 mmol/L
* Medications known to lower the seizure threshold must be discontinued or substituted at least 4 weeks prior to day 1 of study
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug
* Ability to understand, and the willingness to sign, a written informed consent document, as well as comply with study requirements

Exclusion Criteria:

* Subjects who are unwilling to stop taking saw palmetto, PC-SPECs or other herbal agents known to affect the PSA
* Patients may not have received any other investigational agents within 30 days prior to day 1 of study
* Prior exposure to apalutamide, enzalutamide, abiraterone acetate, darolutamide, or any other second-generation antiandrogen therapy

  * Note: prior exposure to bicalutamide, flutamide, nilutamide, or any other first-generation androgen receptor antagonist is permitted. No washout is required. Subjects may be on one of these at the time of consent, but it must be stopped prior to day 1 of study treatment. These drugs are frequently used in the newly diagnosed metastatic setting to blunt the effect of the testosterone spike
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to apalutamide or other agents used in the study
* Subject has another active malignancy other than non-melanomatous skin cancer (unless it is metastatic) or superficial bladder cancer
* Either of the following:

  * Seizure or known condition that may pre-dispose to seizure (e.g. prior stroke within 1 year, brain arteriovenous malformation, Schwannoma, meningioma, or other benign central nervous system [CNS] or meningeal disease which may require treatment with surgery or radiation therapy)
  * Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure or left ventricular ejection fraction < 50%, arterial or venous thromboembolic events (e.g. pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to day 1 of study
* Current evidence of any of the following:

  * Uncontrolled hypertension
  * Gastrointestinal disorder affecting absorption
  * Active infection (e.g. human immunodeficiency virus [HIV] or viral hepatitis)
  * Any chronic medical condition requiring a higher dose of corticosteroid than a total of 10 mg prednisone/prednisolone daily
  * Any condition that in the opinion of the investigator, would preclude participation in this study.
  * Avoid concomitant strong CYP3A4 inducers during abiraterone acetate treatment. If a strong CYP3A4 inducer must be co-administered, increase the abiraterone acetate dosing frequency to twice a day only during the co-administration period (e.g., from 1,000 mg once daily to 1,000 mg twice a day).
  * Avoid co-administration of abiraterone acetate with CYP2D6 substrates that have a narrow therapeutic index. If an alternative treatment cannot be used, exercise caution and consider a dose reduction of the concomitant CYP2D6 substrate
  * Baseline moderate and severe hepatic impairment (Child Pugh Class B & C)
* Inability to stop a prohibited medication:

  * Atypical antipsychotics (e.g. clozapine, olanzapine, risperidone, ziprasidone)
  * Bupropion
  * Lithium
  * Meperidine and pethidine
  * Phenothiazine antipsychotics (e.g. chlorpromazine, mesoridazine, thioridazine)
  * Tricyclic antidepressants (e.g. amitriptyline, desipramine, doxepin, imipramine, maprotiline, mirtazapine
  * Tramadol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Complete prostate specific antigen (PSA) response | At 12 months from the start of treatment
  The complete PSA response is defined as a PSA =< 0.2 ng/ml, confirmed with a 2nd measurement at least 3 weeks later. The estimated PSA response rate will be computed with 95% exact confidence interval. Binomial exact test will be used to determine whether the complete PSA response rate is significantly greater than 43%.

SECONDARY OUTCOMES:
Overall survival | From day 1 of treatment, assessed up to 10 years
  Overall survival will be assessed with each patient visit. After the subject is off active follow up, survival will be assessed by phone.
Incidence of adverse events >= grade 2 | Up to 10 years
  Determined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Proportion of patients with PSA response >= 50% decrease | From baseline, assessed up to 12 months
  The proportion will be reported with 95% confidence interval.
Proportion of patients with PSA response >= 90% decrease | From baseline, assessed up to 12 months
  The proportion will be reported with 95% confidence interval.
Time to treatment failure | From start of treatment, assessed up to 10 years
  Kaplan-Meier plot will be used to describe the survival distributions.
Time to biochemical (PSA) progression | From start of treatment, assessed up to 10 years
  Kaplan-Meier plot will be used to describe the survival distributions.
Time to radiographic progression | From start of treatment, assessed up to 10 years
  Kaplan-Meier plot will be used to describe the survival distributions.
Time to symptomatic progressive disease | From start of treatment, assessed up to 10 years
  Kaplan-Meier plot will be used to describe the survival distributions.
Time to next therapy for metastatic castration resistant prostate cancer | From start of treatment, assessed up to 10 years
  Kaplan-Meier plot will be used to describe the survival distributions.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Graff, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States